CLINICAL TRIAL: NCT06667505
Title: To Co-develop and Test an eHealth Intervention to Improve Knowledge, Attitude and Experience in Patients Living With an Implantable Cardioverter Defibrillator
Brief Title: To Test an e-Health Educational Intervention Patients With an ICD
Acronym: CHOICE-ICD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulster (Other)
Collaborators: Belfast Health and Social Care Trust (Other); Golden Jubilee National Hospital (Other Government)
Responsible Party: Principal Investigator, Loreena Hill, Principal Investigator, University of Ulster
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 24/NI/0094; FS/CDRF/22/21048 (Other Grant/Funding Number: British Heart Foundation)
Record Dates: First submitted 2024-10-11; First posted 2024-10-31 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2024-11

CONDITIONS: Implantable Cardioverter Defibrillator (ICD)
Keywords: Implantable cardioverter defibrillatior; e-Health intervention; patient education

STUDY DESIGN:
Intervention Model Description: Patients, meeting the inclusion criteria of either awaiting or with a recently implanted ICD, will be invited to participate by a member of the clinical team in Belfast Health and Social care Trust (BHSCT) or Golden Jubilee National Hospital (Clydebank). If the patient is interested in participating, they will be invited to nominate a family member.
  Once patients and family member / caregiver provides written informed consent will be randomly allocated to receive the intervention (Choice ICD APP and BHF booklet) or usual care.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CHOICE-ICD (Active Comparator): Patients will receive access to the CHOICE-ICD App for 3 months. They will also be provided with the information booklet, similar to usual care group
  Interventions: Behavioral: Choice-ICD
- Control (No Intervention): Patients will receive information booklet, that they would have received if they had not been included in this research

INTERVENTIONS:
Behavioral: Choice-ICD — The eHealth intervention theoretically driven, interactive and provides personalised information to patients and family members when and where they wish to access it. Five short (2-3 minutes) videos, involving patients, caregivers and professionals, are uploaded onto the APP, alongside animation clips and useful links to online resources. A discussion forum will be accessible for participants using the APP, which will be closely moderated by the researcher, who will ensure any concerning posts or dialogue are promptly removed, and the necessary action is taken. The diary function will allow patients to record and be reminded of future appointments. Patients and family members will engage with the intervention for 3 months.
  Arms: CHOICE-ICD

SUMMARY:
Role of the implantable cardioverter defibrillator (ICD) is to monitor heart rate and discharge a small electrical discharge or shock if the heart rate becomes life threatening. Patients and family members have requested more information about their ICD, how it works and how to live well with the device. This study will build on previous research by designing, in collaboration with patients, family members and professionals, an online resource to provide important information that can lower anxiety and concerns, and improve quality of life. The CHOICE-ICD resource will be easy to use, incorporating games and quizzes to encourage engagement, up to date information appropriate to each patient's needs, as well as animation clips, virtual reality, and short patient videos. CHOICE-ICD will be made available to 64 patients, in addition to normal care, awaiting or with a recently implanted ICD in Belfast and Glasgow. Patients will use the resource for 3 months. Patients and family members will then be asked to complete questionnaires and participate in semi-structured interviews. This study will develop 1st UK online resource providing information to enable patients to have greater choice and control in their care.

DETAILED DESCRIPTION:
Implantable cardioverter defibrillator (ICD) is cornerstone in treatment of life-threatening arrhythmias, yet 25% of patients express concerns following implantation.

Aim: To co-design, optimize and establish feasibility and acceptability of eHealth intervention: CHOICE-ICD, providing information to reduce patients' concerns and improve quality of life.

Methods: Phase 1 has been completed: Underpinned by theory and research, core components of an intervention has been co-designed according to six-step process, and in collaboration with stakeholders. Components include ICD written information, educational animations, virtual reality application and patient videos. International advisory group will oversee iterative development, user testing and optimization.

Phase 2 ongoing: CHOICE-ICD is pilot trial, recruiting 128 patients awaiting/recently implanted ICD or cardiac resynchronisation therapy with ICD from Northern Ireland and Glasgow. Participants will use the intervention for 3 months. Data will be analyzed to determine feasibility and acceptability of intervention, and trial methods for future effectiveness trial.

Outcomes: Recruitment, consent and randomization rates, and completion of questionnaires at baseline, 3 and 6 months. Acceptability of intervention delivery and suitability of outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Patients with heart failure awaiting or with an ICD (no time restriction on implantation)
* No cognitive impairment

Caregivers:

* Have contact with the patient at least 5 times per week.
* Be physically and mentally capable of participation (self-assessment)

Healthcare professionals:

* Daily care of patients with heart failure and an implantable cardioverter defibrillator
* Involved in the care of a patient using the Choice-ICD intervention

Exclusion Criteria:

* Patients, judged by their Cardiologist as physically or mentally unsuitable to complete the study.
* Patients or caregivers lacking capacity to give consent.
* Patients who have known pregnancy
* Caregivers who's patient is unwilling to take participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility, acceptability and usability of the Choice-ICD intervention | 3 and 6 months after recruitment.
  System Usability Scale and focus group. The system usability scale has 10 questions, with responses on a Likert scale 1(strongly disagree) to 5 (strongly agree). The higher the score the more feasible. The focus group will be completed at 6 months.

SECONDARY OUTCOMES:
Patients' perceptions pre and post intervention | Baseline, 3 months and 6 months.
  Brief Illness perception questionnaire. The Brief Illness questionnaire has 8 questions, with responses on a Likert scale 1 to 10 Likert Scale (the higher the score (maximum 30) the more positive the patient's view.
Patients' concerns regarding the ICD pre and post intervention | Baseline, 3 months and 6 months.
  Implantable Cardioverter Defibrillator concerns questionnaire (ICDC).The validated questionnaire has 20 questions, with responses ranging from not at all to very much. The more worried the patient is, the higher the score ( maximum 100).
Patients' knowledge, experience and attitudes pre and post intervention | Baseline, 3 months and 6 months.
  Experiences, Attitudes and Knowledge of End-of-Life issues in Implantable Cardioverter Defibrillator Questionnaire (EOL-ICDQ). Validated questionnaire with 17 questions, the higher the score indicates the lower level of knowledge on the device
Patients' anxiety pre and post intervention | Baseline, 3 months and 6 months.
  Beck Anxiety Inventory (BAI). Validated questionnaire with 21 questions, with responses from "not at all anxious" to "severely anxious", therefore the higher the scoring the more anxiety.
Patients' acceptance of the ICD pre and post intervention | Baseline, 3 months and 6 months.
  Florida Patient Acceptance Survey (FPAS). Validated questionnaire with 18 questions, responses on a Likert scale of 1-5, with lower score indicating higher level of acceptance of device
Patients' quality of life pre and post intervention | Baseline, 3 months and 6 months.
  Kansas City Cardiomyopathy questionnaire (KCCQ- 12) quality of life tool. Validated questionnaire with 8 key questions, scores are 0-100, where 0 notes lowest health status and 100 highest possible health status
Caregiver burden pre and post intervention | Baseline, 3 months and 6 months.
  Carer Strain Index (CSI). Validated questionnaire with 12 questions and responses as Yes or No. A score of 7 or higher indicates a high level of stress.

CONTACTS AND LOCATIONS:
Overall Officials: Loreena M Hill, PhD, Principal Investigator — Ulster University

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2024-07-30): https://cdn.clinicaltrials.gov/large-docs/05/NCT06667505/Prot_000.pdf